CLINICAL TRIAL: NCT04136990
Title: Comparison of Anterior Cruciate Ligament Isolated Reconstruction or Combined With Lateral Extra-articular Tenodesis in Knee Laxity, Graft Failure and Patient-reported Outcome Measures
Brief Title: Does ACL Augmented With LEAT Better Controls Rotational Laxity Than Isolated ACL Reconstruction?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Espregueira-Mendes Sports Centre - FIFA Medical Centre of Excellence (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0015/0019
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: Anterior Cruciate Ligament Reconstruction; Lateral Extra-Articular Tenodesis; Knee Laxity; Porto Knee Testing Device
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Non-randomized 1:1 allocation
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blinded to the patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated ACL reconstruction (Active Comparator): Isolated ACL reconstruction only.
  Interventions: Procedure: Isolated ACL reconstruction
- ACL + LEAT (Experimental): ACL reconstruction combined with Lateral Extra-Articular Tenodesis (LEAT).
  Interventions: Procedure: ACL + LEAT reconstruction

INTERVENTIONS:
Procedure: Isolated ACL reconstruction — Isolated ACL reconstruction using the bone-patellar tendon autograft.
  Arms: Isolated ACL reconstruction
Procedure: ACL + LEAT reconstruction — ACL reconstruction using the bone-patella-tendon-bone autograft combined with LEAT using the mini Lemaire technique.
  Arms: ACL + LEAT

SUMMARY:
It has been suggested that adding a Lateral Extra-Articular Tenodesis (LEAT) to Anterior Cruciate Ligament (ACL) reconstruction has the advantage of better controlling the rotational laxity. The objective of this study is to compare the the sagittal and rotational knee laxity using the Porto Knee Testing Device (PKTD) - a MRI-compatible arthrometer - at 2 years follow-up (side-to-side and to baseline comparison) in patients that underwent isolated ACL reconstruction (isolated ACL) versus ACL reconstruction combined with LEAT (ACL+LEAT). Patient-reported outcome measures using the Knee Injury and Osteoarthritis Outcome Score (KOOS) and graft failure (re-tear) will also be assessed at 2 years follow-up.

DETAILED DESCRIPTION:
This study is a non-randomized clinical trial including 40 patients with anterior cruciate ligament injury who are undergoing surgery and will be allocated 1:1 to either isolated ACL reconstruction (control group) or ACL reconstruction combined with lateral extra-articular tenodesis (experimental group). The principal outcome of this work is the sagittal and rotational knee laxity analysis and side-to-side and 2-year improvement. The secondary outcomes include graft failure (re-tears) and the patient-reported outcome measures (KOOS) at 2 years follow-up.

ELIGIBILITY:
Inclusion Criteria:

* no previous knee surgeries
* contralateral healthy knee
* positive pivot-shift (++)

Exclusion Criteria:

* revision ACL surgery
* ACL reconstruction using allograft or synthetic grafts
* multi-ligament injury
* pregnant female
* other injuries or conditions that may alter the knee function (eg. severe osteoarthritis)
* requiring concomitant osteotomy
* requiring concomitant cartilage surgery (other than debridement)

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of sagittal and rotational knee laxity | Baseline and 24 months
  To assess the post-operative knee sagittal and rotational laxity, we will use the Porto Knee Testing Device (PKTD). We will measure the anterior displacement on the medial and lateral plateaus and internal and external rotation in the lateral and medial plateau. Additionally, these measures will be combined to measure the anterior global translation (anterior translation on lateral + medial plateaus) and the global rotation (internal + external rotation in the lateral plateau).

SECONDARY OUTCOMES:
Graft Failure | 24 months
  Rate of graft failure. It will be considered only graft tears. We will determine the absolute risk of graft failure in each group, if enough data available.
Change from baseline of Knee Osteoarthritis and Outcomes Score (KOOS) | Baseline, 12 and 24 months
  The KOOS is a 42-item knee-specific questionnaire with five separately reported domains, including pain (9 items), other symptoms (7 items), function in daily living (17 items), function in sports/recreation (5 items) and knee-related quality of life (4 items). Domain scores represent the average of all items in the domain standardized to a score from 0 to 100 (worst to best).
Change from baseline of Tegner Scale | Baseline, 12 and 24 months
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10, developed for knee injuries (especially ACL injury).

CONTACTS AND LOCATIONS:
Overall Officials: João Espregueira-Mendes, MD, PhD, Study Director — Clínica do Dragão, Espregueira-Mendes Sports Centre - FIFA Medical Centre of Excellence; Renato Andrade, Principal Investigator — Clínica do Dragão, Espregueira-Mendes Sports Centre - FIFA Medical Centre of Excellence
Locations (1):
- Clínica do Dragão, Espregueira-Mendes Sports Centre - FIFA Medical Centre of Excellence, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No